CLINICAL TRIAL: NCT01060826
Title: Randomized, Double-blind Study to Evaluate the Efficacy of Administration With Intravenous Bolus Followed by a Continuous Infusion of Somatostatin in the Prevention of Post-ERCP Pancreatitis
Brief Title: Efficacy of Administration of Somatostatin in the Prevention of Post-endoscopic Retrograde Cholangiopancreatography (ERCP) Pancreatitis
Acronym: crepsmt1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Cristina Gómez Oliva (principal investigator), Cristina Gómez
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2008-003338-41; 2008-003338-41 (EudraCT Number)
Record Dates: First submitted 2010-01-28; First posted 2010-02-02 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Acute Pancreatitis
Keywords: acute pancreatits
MeSH Terms: conditions — Pancreatitis | interventions — Somatostatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- somatostatin, intravenous bolus (Experimental): A double- blind study designed to evaluate if the treatment with somatostatin in intravenous bolus before starting the ERCP procedure followed by a continuous infusion for 4 hours after endoscopic proof could prevent acute post-ERCP pancreatitis. Patients submitted to ERCP will be randomized in two groups of treatment, one will receive somatostatin and another placebo.
  Interventions: Drug: somatostatin, intravenous bolus; Drug: somatostatin
- Placebo, intravenous bolus (Placebo Comparator): A double- blind study designed to evaluate if the treatment with somatostatin in intravenous bolus before starting the ERCP procedure followed by a continuous infusion for 4 hours after endoscopic proof could prevent acute post-ERCP pancreatitis. Patients submitted to ERCP will be randomized in two groups of treatment, one will receive somatostatin and another placebo.
  Interventions: Other: fisiologic serum

INTERVENTIONS:
Other: fisiologic serum — 250 microgramos bolus intravenous during 3 minutes and continuous infusion for 4 hours after endoscopic procedure
  Arms: Placebo, intravenous bolus
Drug: somatostatin, intravenous bolus — 250 microgramos bolus intravenous in 3 minutes and continuous infusion for 4 hours after endoscopic
  Arms: somatostatin, intravenous bolus
Drug: somatostatin — Intravenous bolus 250 micrograms
  Arms: somatostatin, intravenous bolus

SUMMARY:
Acute pancreatitis is the most frequent (5-10%) and severe complication after endoscopic retrograde cholangiopancreatography (ERCP), that could require of surgical intervention and lead to death. A double- blind study designed to evaluate if the treatment with somatostatin in intravenous bolus before starting the ERCP procedure followed by a continuous infusion for 4 hours after endoscopic proof could prevent acute post-ERCP pancreatitis. Patients submitted to ERCP will be randomized in two groups of treatment, one will receive somatostatin and another placebo. The main aim of this study will be the incidence of acute post-ERCP pancreatitis and secondary objectives will be identify sub-groups of patient with high risk to develop post-ERCP pancreatitis, who could benefit of pharmacologic prophylaxis before the exploration. The study will include 510 patients submitted to an ERCP during a period of 3 years.

DETAILED DESCRIPTION:
A double- blind study designed to evaluate if the treatment with somatostatin in intravenous bolus before starting the ERCP procedure followed by a continuous infusion for 4 hours after endoscopic proof could prevent acute post-ERCP pancreatitis. Patients submitted to ERCP will be randomized in two groups of treatment, one will receive somatostatin and another placebo. The main aim of this study will be the incidence of acute post-ERCP pancreatitis and secondary objectives will be identify sub-groups of patient with high risk to develop post-ERCP pancreatitis, who could benefit of pharmacologic prophylaxis before the exploration. The study will include 510 patients submitted to an ERCP during a period of 3 years.

ELIGIBILITY:
Inclusion criteria:

1. Patients undergoing therapeutic endoscopic retrograde cholangiopancreatography (ERCP).

Exclusion Criteria:

1. Pregnancy or history of allergy to somatostatin.
2. Acute myocardial infarction within 3 months of the procedure.
3. Acute pancreatitis in patients undergoing early ERCP in the acute phase of the disease.
4. Previous sphincterotomy.
5. Chronic pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
The incidence of acute post-ERCP pancreatitis | One week

SECONDARY OUTCOMES:
Identify sub-groups of patients with high risk to develop post-ERCP pancreatitis | One week

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Gómez, Principal Investigator — Endoscopy Unit
Locations (2):
- Spain (2):
  - Endoscopy Unit Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona

REFERENCES:
- [Background] 1. Cotton PB, Lehman G, Vennes J, et al. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc 1991;37:383-93. 2. Freeman ML, Guda NM. Prevention of post-ERCP pancreatitis: a comprehensive review. Gastrointest Endosc 2004;59:845-64. 3. Bordás JM et al. Effects of bolus somatostatin in preventing pancreatitis after endoscopic pancreatography: results of a randomized study. Gastrointest Endosc 1998;47:230-4. 4. Poon RT, Yeung C, Liu CL, et al. Intravenous bolus somatostatin after diagnostic cholangiopancreatography reduces the incidence of pancreatitis associated with therapeutic endoscopic retrograde cholangiopancreatography procedures: a randomized controlled trial. Gut 2003;52:1768-73. 5. Andriulli A et al. Pharmacologic treatment can prevent pancreatic injury after ERCP: a meta-analysis. Gastrointest Endosc. 2000;5:1-7.
- [Derived] Concepcion-Martin M, Gomez-Oliva C, Juanes A, Diez X, Prieto-Alhambra D, Torras X, Sainz S, Villanueva C, Farre A, Guarner-Argente C, Guarner C. Somatostatin for prevention of post-ERCP pancreatitis: a randomized, double-blind trial. Endoscopy. 2014 Oct;46(10):851-6. doi: 10.1055/s-0034-1377306. Epub 2014 Jun 30. PMID 24977398
- See also: preventing post-therapeutic ERCP pancreatitis — http://www.gastro.org